CLINICAL TRIAL: NCT03339791
Title: Sleeve Gastrectomy Versus Roux-en-Y Gastric Bypass for Treatment of Severe Obesity in Patients With 65 Years or Older: a Randomized Controlled Trial - The "BaSE" Trial - Bariatric Surgery in the Elderly.
Brief Title: Sleeve Versus Bypass in Older Patients: a Randomized Controlled Trial
Acronym: BaSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Denis Pajecki, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 68401117.4.0000.0068
Record Dates: First submitted 2017-10-30; First posted 2017-11-13 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Obesity, Morbid; Surgery; Elderly
MeSH Terms: conditions — Obesity, Morbid | interventions — Gastric Bypass

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleeve (Active Comparator): Morbid obese patients, 65 years old or more, submitted to Sleeve Gastrectomy
  Interventions: Procedure: Sleeve Gastrectomy
- Bypass (Active Comparator): Morbid obese patients, 65 years old or more, submitted to Gastric Bypass
  Interventions: Procedure: Gastric Bypass

INTERVENTIONS:
Procedure: Sleeve Gastrectomy — Laparoscopic Sleeve Gastrectomy. Technique: complete mobilization of the greater curvature and gastric fundus up to the angle of Hiss; stapling beginning at 3 to 4 cm away from the pylorus; bougie size 32 French; oversuture of the staple line; hiatoplasty in selected cases; routine drainage of the abdominal cavity
  Other Names: Vertical gastrectomy
  Arms: Sleeve
Procedure: Gastric Bypass — Laparoscopic Gastric Bypass. Technique: Pouch size 30 to 40 ml, biliopancreatic limb 70 to 100 cm, alimentary limb 100 to 120 cm, antecolic, routine closure of the mesenterial defects, routine drainage of the abdominal cavity
  Other Names: Roux-en_y Gastric Bypass
  Arms: Bypass

SUMMARY:
The aim of the study is to compare two different bariatric procedures performed in patients with 65 years or more: gastric bypass and sleeve gastrectomy. Primary outcomes will be weight loss, control of comorbidities and morbidity of the operation. Secondary outcomes are related to functionality, that will be evaluated with specific tests.

DETAILED DESCRIPTION:
Introduction: Surgical treatment of obesity in patients over 65 years of age is controversial. For patients in this age group, there is a prevailing concept that the risk / benefit ratio of the procedure should be evaluated for each individual patient, without determining objective criteria or outcomes that characterize this benefit. Increased surgical risk in patients older than 65 years is undoubtedly a limiting factor for the broader indication of bariatric surgery in this population. The two most applied surgical techniques are Sleeve Gastrectomy and Roux-en-Y Gastric Bypass. Most of the studies that evaluated the two techniques in elderly patients are retrospective, prospective non-randomized, or contemplated only one technique. Recent, studies concluded that in the elderly the weight loss with Gastric Bypass was higher, but the surgical morbidity with the Sleeve was lower and there was no difference in the resolution of comorbidities between the two techniques. In evaluating the benefits of surgery, most studies address outcomes such as weight loss and control of metabolic and cardiovascular comorbidities. Outcomes that are specific to the treatment of obesity in the elderly, such as improvement of functionality, decreased fragility and improvement of the quality of life have not been studied yet. In this field, there is concern that excessive weight loss, accompanied by loss of muscle mass may compromise the mentioned parameters, especially in individuals who already have loss of bone and muscle mass before surgery. For this reason, the assessment of bone mass and body composition in the preoperative period of these individuals is fundamental. In order to identify the benefits of weight loss promoted by surgery and life expectancy, the elderly patients in preparation for operation at the Bariatric Surgery Unit of the Hospital das Clinicas University of São Paulo School of Medicine are submitted to a geriatric evaluation, which includes the analysis of their functional dependency profile, Important prognostic factor in this population. Objectives: The primary objective of the study will be to evaluate surgical morbidity and short-term (weight loss, comorbid control) outcomes of surgical treatment of obesity in patients over 65 years of age, comparing two techniques: Sleeve Gastrectomy (SG) and Gastric Bypass (GB). The secondary objective will be to evaluate the body composition of the individuals, before and after the surgery, comparing the two techniques. Patients and methods: This is a prospective study, in which 40 consecutive patients, aged 65 years and over, will be admitted to the Bariatric and Metabolic Surgery Unit of the Discipline of Digestive System Surgery of Hospital das Clinicas University of São Paulo School of Medicine with indication criteria for bariatric surgery. Patients will be randomized into two groups according to the surgical technique to be used: SG or GB. Data related to surgical morbidity, weight loss, control of comorbidities, nutritional deficiencies, changes in body composition and functionality will be evaluated and compared after a follow-up of at least 12 months.

ELIGIBILITY:
Inclusion Criteria:

* BMI over 40 Kg/m2 for at least 5 years with failure of obesity medical treatments
* BMI over 35 Kg/m2 with at least 2 comorbidities and failure of medical treatments

Exclusion Criteria:

* prior bariatric surgery
* clinical or psychological conditions that contraindicate bariatric surgery

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-09-23 (Actual); Primary Completion 2017-11-07 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Total Weight loss | 1 year
  Weight loss measured in percentage of weight loss (%WL)
Surgical Complications | 30 days
  Bleeding, Leakage, Fistula, Bowel obstruction
Mortality | 90 days
  mortality
Improvement of Type II diabetes | baseline and 1 year
  Measure of glycated hemoglobin
Improvement of hypertension | baseline and 1 year
  measure of blood pressure (mmHg)
Improvement of LDL | baseline and 1 year
  measure of LDL
Clinical complications | 30 days
  cardiac, pulmonary, other
Excess weight loss | 1 year
  excess weight loss (%EWL); considering the normal weight the equivalent to the BMI 25 Kg/m2
Improvement of hypertension by use of medication | baseline and 1 year
  evaluation of the number of drugs used to treat hypertension
Improvement of HDL | baseline and 1 year
  measure of HDL
Improvement of triglycerides | baseline and 1 year
  measure of triglycerides

SECONDARY OUTCOMES:
Functionality | baseline and 1 year
  Functionality specific test (Activities of Day living)
Body composition | baseline and 1 year
  Dexa (Dual-energy X-ray absorptiometry) body composition study
Functionality | baseline and 1 year
  Functionality specific test (Instrumental activities of day living)
Functionality | baseline and 1 year
  Time up and go test

CONTACTS AND LOCATIONS:
Overall Officials: Denis Pajecki, Principal Investigator — Hospital das Clinicas - Faculdade de Medicina da USP
Locations (1):
- Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The plan is to publish the complete data after the end of the study

REFERENCES:
- [Background] Maghrabi AH, Wolski K, Abood B, Licata A, Pothier C, Bhatt DL, Nissen S, Brethauer SA, Kirwan JP, Schauer PR, Kashyap SR. Two-year outcomes on bone density and fracture incidence in patients with T2DM randomized to bariatric surgery versus intensive medical therapy. Obesity (Silver Spring). 2015 Dec;23(12):2344-8. doi: 10.1002/oby.21150. Epub 2015 Jul 20. PMID 26193177
- [Background] Abbas M, Cumella L, Zhang Y, Choi J, Vemulapalli P, Melvin WS, Camacho D. Outcomes of Laparoscopic Sleeve Gastrectomy and Roux-en-Y Gastric Bypass in Patients Older than 60. Obes Surg. 2015 Dec;25(12):2251-6. doi: 10.1007/s11695-015-1712-9. PMID 26001882
- [Background] Pajecki D, Santo MA, Kanagi AL, Riccioppo D, de Cleva R, Cecconello I. Functional assessment of older obese patients candidates for bariatric surgery. Arq Gastroenterol. 2014 Jan-Mar;51(1):25-8. doi: 10.1590/s0004-28032014000100006. PMID 24760060
- [Background] Strain GW, Gagner M, Pomp A, Dakin G, Inabnet WB, Saif T. Comparison of fat-free mass in super obesity (BMI >/= 50 kg/m2) and morbid obesity (BMI <50 kg/m2) in response to different weight loss surgeries. Surg Obes Relat Dis. 2012 May-Jun;8(3):255-9. doi: 10.1016/j.soard.2011.09.028. Epub 2011 Oct 20. PMID 22118843